CLINICAL TRIAL: NCT00431522
Title: Protective Effect of Valproate on Brain Cells:A Magnetic Resonance Imaging and Spectroscopy Study in Patients With Bipolar Disorder Diagnosis
Brief Title: Valproic Acid Sodium Salt in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: L_9387
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

INTERVENTIONS:
Drug: Valproic acid, sodium salt

SUMMARY:
* To determine the total and local gray matter volumes, and N-acetyl aspartate (NAA) levels in patients with bipolar disorders who are within euthimic, depressive or manic/hypomanic period and who are not taking drug;
* To investigate the neuroprotective effects of long-term (6 weeks) use of valproate on total and local gray matter volumes and NAA levels.
* To measure the brain electrical response to visual and auditory impulses before and after valproate treatment in patients within euthimic, depressive or manic/hypomanic period and who are not taking drug, and to compare the data with each other and with normal groups.
* To determine the cognitive functions before and after the valproate treatment in the same patient group, to compare the data with each other and with age- and sex-paired normal controls;
* To determine the relationship between these effects of valproate and clinical improvement;
* To investigate the relationship between cognitive ability status and electrical activity of brain, to compare this with that in control group; to determine the relationship between the data and brain imaging (MRI/MRS) findings in conjunction with localization

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type I or II bipolar disorder according to DSM-IV after stratified SCID I interview,
* being currently euthimic (for at least one month), manic-hypomanic and having YMRS points of 15 or more, or being in depressive episode and having HAM-D21 points of 15 or more
* being not taking drugs for at least two weeks before participating in the study (except benzodiazepins)

Exclusion Criteria:

* female who are pregnant or planning to be pregnant, nursing
* having known hypersensitivity to study drug
* being given any psychotropic agent other than benzodiazepine within the last two weeks
* active sustance or alcohol usage within the last two weeks, or substance addiction other than cafein or nicotine (within the last month)
* having another axis I disorder such as comorbid dementia, delirium, obsessive compulsive disorder, eating disorder
* having unstabilised hepatic or renal disorder, thyroid or blood disease
* having history of cerebral surgery
* existence of a degenerative neurologic disease or epilepsy
* having pacemaker
* having a prosthesis able to magnetic effect in eye, brain or sites near to these regions
* homicide thougths or severe catatonia required to be hospitalized
* having mixed episode

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-12; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To assess regional N-acetyl aspartate (NAA) levels in drug free bipolar patients either in manic/hypomanic, or depressive or euthymic state | for 6 weeks
To investigate valporate's effect on total and regional gray matter volume and NAA levels; | for 6 weeks

SECONDARY OUTCOMES:
To assess evoked and event related potentials to visual and auditory stimuli in patients before and after valproate monotherapy in comparison to healthy controls | for 6 weeks
To determine the relationship between clinical improvement and image data changes in depressed or manic/hypomanic patients, | for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edibe Taylan, Study Director — Sanofi-aventis Turkey
Locations (1):
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)